CLINICAL TRIAL: NCT04292067
Title: Characterisation of Intestinal Microbiota of Patients With Spondyloarthritis or Rheumatoid Arthritis
Acronym: MICROBIART
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190991; 2019-A02632-55 (Registry Identifier: IDRCB)
Record Dates: First submitted 2020-02-26; First posted 2020-03-02 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-05

CONDITIONS: Spondyloarthritis; Rheumatoid Arthritis
Keywords: Spondyloarthritis; Rheumatoid Arthritis; Microbiota
MeSH Terms: conditions — Spondylarthritis; Arthritis, Rheumatoid | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Faecal sampling at baseline for each subject
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- patients with SPA: 100 SPA patients
  Interventions: Biological: Faecal sampling; Biological: Blood sampling
- Healthy subjets: 200 healthy subjets in control group
  Interventions: Biological: Faecal sampling; Biological: Blood sampling
- patients with RA: 100 RA patients
  Interventions: Biological: Faecal sampling; Biological: Blood sampling

INTERVENTIONS:
Biological: Faecal sampling — Faecal sampling at baseline
Biological: Blood sampling — Blood sampling at baseline

SUMMARY:
The primary objective of the study aims to compare the biodiversity of intestinal microbiota between spondylarthritis (SPA) or rheumatoid arthritis (RA) patients and healthy volunteers, by microbiota DNA sequencing in order to further and respond the prior results, which suggested that there is a specific dysbiosis for each of the 2 diseases. A comparative analysis will allow to identify the biomarkers of the specific bacteria.

DETAILED DESCRIPTION:
As secondary objectives, the study aims to analyse the relation between different clinical parameters such as age, gender, duration of the disease, or the nature of ongoing treatment, and the the composition of intestinal microbiota, and identify dysbiosis of bacteria, which will be specific functional signatures of intestinal microbiota in SPA and/or RA. Analyse the relation between metabolome of faecale and plasma and the composition of intestinal microbiota.

This study will be performed in the rheumatology department in Ambroise Paré hospital of APHP group in France.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Patient ⩾ 18 years;
* Diagnosed as spondyloarthritis (SpA) according ASAS classification, or rheumatoid polyarthritis according ACR/EULAR;
* Affiliated to a social security scheme;
* Have signed the written informed consent form.

Healthy control subjects:

* Adult women and men;
* Subjet free of chronic pathology;
* Affiliated to a social security scheme;
* Have signed the written informed consent form.

Exclusion Criteria:

Patients:

* Patients unable to understand the proposed study and/or sign a informed consent form;
* Pregnant women or breast feeding women;
* Patient ⩾ 18 years;
* Patients under guardianship or curatorship;
* Have taken antibiotic 1 month prior to inclusion or digestive coloscopy 6 months prior inclusion;
* Presenting acute or chronic severe pathology may likely to interfere with the interpret of outcome;
* Foreign patients under french AME scheme;
* Patients had have participated in the prior study Microbiart.

Healthy control subjects:

* Subjects unable to understand the proposed study and/or sign a informed consent form;
* Pregnant women or breast feeding women;
* Subjects < 18 years;
* Subjects under guardianship or curatorship;
* Presenting acute or chronic severe pathology may likely to interfere with the interpret of outcome;
* Refusal of subjects to participate to the study;
* Foreign patients under french AME scheme;
* Subjects had have participated in the prior study Microbiart.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Adult patient diagnosed spondyloarthritis or rheumatoid polyarthritis;
  * Healthy adult subjects free of chronic pathology.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-11-23 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Bacteria analysis | At the end of study, up to 4 years
  Quantitative analysis of repartition of bacteria in each group and the comparison between groups.

SECONDARY OUTCOMES:
Intestinal microbiota composition | At the end of study, up to 4 years
  Intestinal microbiota composition will be analysed

CONTACTS AND LOCATIONS:
Overall Officials: Maxime BREBAN, MD, PhD, Principal Investigator — Service de Rhumatologie, Hôpital Ambroise Paré, APHP
Locations (1):
- Service de Rhumatologie, Hôpital Ambroise Paré, Assistance Publique-Hôpitaux de Paris, Boulogne-Billancourt, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Breban M, Tap J, Leboime A, Said-Nahal R, Langella P, Chiocchia G, Furet JP, Sokol H. Faecal microbiota study reveals specific dysbiosis in spondyloarthritis. Ann Rheum Dis. 2017 Sep;76(9):1614-1622. doi: 10.1136/annrheumdis-2016-211064. Epub 2017 Jun 12. PMID 28606969